CLINICAL TRIAL: NCT06891170
Title: B Cell Responses in COVID-19: Generation of SARS-CoV-2 Neutralizing Human Monoclonal Antibodies to Efficiently Contrast Wild-type and Emerging Variants.
Brief Title: B Cell Responses in COVID-19
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Barbara Oliviero, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: RC_08072721
Record Dates: First submitted 2025-03-21; First posted 2025-03-24 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-03

CONDITIONS: COVID 19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Vaccinated or recovered subjects from COVID-19

SUMMARY:
In this study, we will develop techniques to optimize the in vitro production of human monoclonal antibodies.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 at time of signing informed consent form
* Signed informed consent form

Exclusion Criteria:

* Ongoing drug abuse
* Active or history of neoplastic malignancy
* Active autoimmune disease ongoing treatment with immunosuppressive therapy
* Ischemic heart disease
* Evidence of positive HIV, HCV, HBV test
* Diabetes
* Failure to sign informed consent form

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Vaccinated or recovered subjects from COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Optimization of the method to obtain human mAbs neutralizing COVID-19. | From enrollment to 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia, Pavia, Italy